CLINICAL TRIAL: NCT01638520
Title: Safety and Efficacy of Blocking IL-4 With Pascolizumab in Patients Receiving Standard Combination Therapy for Pulmonary Tuberculosis (TB): a Randomized, Double-blind, Placebo-controlled, Proof-of-concept Clinical Trial
Brief Title: Safety and Efficacy of Blocking IL-4 With Pascolizumab in Patients Receiving Standard Therapy for Pulmonary Tuberculosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSRB 2012/02212
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Immune Therapy; Interleukin 4; monoclonal antibody
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pascolizumab (Experimental): The dose of study medication will be calculated using the patient's body weight and the appropriate dosing regimen based on the cohort of enrollment. The medication will be administered by slow intravenous infusion over 1 hour under close medical supervision.
  Interventions: Drug: Pascolizumab
- Placebo (Placebo Comparator): For patients randomized to placebo, Sterile 0.9% w/v Sodium Chloride will be used for Injection, using the same volume that would have been prepared if the patient had been randomized to receive pascolizumab.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pascolizumab — 0.05mg/kg - 10mg/kg Pascolizumab according to dosing cohort
  Arms: Pascolizumab
Drug: Placebo — Saline (volume determined based on weight of patient, and cohort of enrollment)
  Arms: Placebo

SUMMARY:
New approaches are needed to achieve more rapid elimination of dormant mycobacteria and thereby shorten treatment for drug-sensitive and drug-resistant tuberculosis (TB). Dormant mycobacteria are relatively resistant to antibacterial drugs and approaches that enhance immune clearance have the potential to be more effective. Interleukin-4 (IL-4) is a key cytokine in the immune response to TB that may impair the clearance of mycobacteria. We hypothesize that pascolizumab, an anti-IL-4 monoclonal antibody, might be of value as an adjunct to standard treatment.

The aims of this trial are to determine whether administration of pascolizumab as an adjunct to standard combination treatment for drug-sensitive TB produces changes in one or more parameters of bacterial or host response (including bacterial clearance, host clinical status, immune response, bacterial and host transcriptomics, lung imaging) that may indicate potential for enhanced sterilization and to confirm the safety of blocking IL-4 (previously demonstrated in healthy volunteers and patients with asthma) in patients with TB.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 -75 years of age
2. Male or female: females eligible only if not of childbearing potential or agree to remain abstinent or use an appropriate contraceptive method during the study.
3. Confirmed pulmonary TB by smear microscopy and Gene Xpert™
4. Absence of rifampicin resistance on molecular probe (Gene Xpert™)
5. Estimated to be able to produce at least 5ml of sputum per 24 hour period.
6. No previous history of anti-TB therapy for active disease (treatment for latent disease acceptable).
7. Willing to comply with the study visits and procedures
8. Willing and able to provide written informed consent

Exclusion Criteria:

1. More than 28 days of standard anti-TB chemotherapy at the time of randomization.
2. Disseminated TB (lymphadenopathy is acceptable)
3. Underlying serious chronic diseases such as those of the liver, kidney disease, blood disorders and Type I diabetes (controlled Type II diabetes is acceptable) or any significant organ dysfunction.
4. History of myocardial infarction, congestive heart failure or arrhythmia within 6 months of screening
5. History or evidence of chronic alcohol consumption or drug abuse
6. Current autoimmune disease or history of autoimmune disease.
7. Known or suspected hypersensitivity to any component of the trial medication (sodium phosphate, sodium chloride, glycine, sucrose, polysorbate 80)
8. Chronic use of an immunosuppressant
9. Treatment with any monoclonal antibody within 6 months of randomization
10. Vaccination within the 6 weeks prior to randomization (patients who have received influenza vaccination can enroll at 2 weeks following vaccination).
11. Seropositive for human immunodeficiency virus-1 or 2; hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at screening
12. Creatinine > 1.4 times upper limit of normal or ALT greater than 2.5 times upper limit of normal on screening blood tests
13. QTc >450 msec on ECG performed at screening
14. Women who are currently pregnant or breastfeeding
15. Any other significant condition that would, in the opinion of the investigator, compromise the patient's safety or outcome in the trial.
16. Participation in other clinical intervention trial or research protocol (Participation in other studies that do not involve an intervention may be allowed, but this must be discussed and approved by Chief Investigator )

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-06; Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy - Time to detection on liquid culture of sputum on Week 8 | 8 weeks post intervention
Co-primary outcome measure - safety | Upto 24 weeks via follow-up visits/assessments and 24-96 weeks via phone assessments
  Adverse events considered at least possibly related to study medication and that are classified by the site investigator as serious and/or grade IV severity

SECONDARY OUTCOMES:
Sputum culture status (positive or negative) on liquid culture at week 8 | 8 weeks
Rate of change (area under the curve) from baseline to week 8 in the time to positivity in liquid culture of sputum | 8 weeks
Rate of change in serial sputum colony counts on solid cultures from baseline to week 8 | 8 weeks
Rate of change of RPF-dependent serial sputum colony counts from baseline to week 8 | 8 weeks
Sputum culture status (positive or negative) on solid culture at week 8 | 8 weeks
Rate of change of sputum smear lipid-body positive mycobacteria from baseline to week 8 | 8 weeks
Serum IL-4 levels (free and drug-bound) | 24 weeks
Time to resolution of fever | 24 weeks
Time to resolution of all TB symptoms | 24 weeks
Resolution of chest X-ray changes at week 24 | 24 weeks
Resolution of PET/MRI changes at week 8 and week 24 | 24 weeks
TB relapse at any time up to week 96 | 96 weeks
Anti-pascolizumab antibodies | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nick Paton, Principal Investigator — National Univesity, Singapore
Locations (7):
- Malaysia (2):
  - Institute of Respiratory Medicine, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Philippines (2):
  - Lung Centre Philippines, Manila
  - Philippines Tuberculosis Society Inc., Manila
- Singapore (3):
  - Changi General Hospital, Singapore
  - National University Hospital, Singapore, Singapore
  - Ng Teng Fong General Hospital, Singapore

REFERENCES:
- [Derived] Paton NI, Gurumurthy M, Lu Q, Leek F, Kwan P, Koh HWL, Molton J, Mortera L, Naval S, Bakar ZA, Pang YK, Lum L, Lim TK, Cross GB, Lekurwale G, Choi H, Au V, Connolly J, Hibberd M, Green JA; Pascolizumab Tuberculosis Trial Team. Adjunctive Pascolizumab in Rifampicin-Susceptible Pulmonary Tuberculosis: Proof-of-Concept, Partially-Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Trial. J Infect Dis. 2024 Sep 23;230(3):590-597. doi: 10.1093/infdis/jiae104. PMID 38527849